CLINICAL TRIAL: NCT06798103
Title: Comparative Study Between Efficacy of Ultrasound-Guided Bilateral Erector Spinae Plane Block and Thoracic Paravertebral Block on Perioperative Analgesia and Fast Recovery of Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Comparing Perioperative Analgesia After Ultrasound Guided Bilateral Erector Spinae Plane Block and Thoracic Paravertebral Block in Laparoscopic Sleeve Gastrectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Ahmed Ahmed, Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD335/2023
Record Dates: First submitted 2025-01-03; First posted 2025-01-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-02

CONDITIONS: Laparoscopic Sleeve Gastrectomy (LSG); Erector Spinae Plane Block; Thoracic Paravertebral Block
Keywords: Laparoscopic Sleeve Gastrectomy (LSG); Erector Spinae Plane Block; Thoracic Paravertebral block

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (ESPB) (Active Comparator): Group (I): 15 participants will be injected with 30 mL of 0.25% bupivacaine deep to the erector spinae muscle.
  Interventions: Procedure: Erector Spinae Plane Block
- Thoracic paravertebral block group (TPVB) (Active Comparator): Group (II): 15 participants will be injected with 25 ml of 0.25% bupivacaine into paravertebral space of T7 vertebra.
  Interventions: Procedure: Thoracic paravertebral block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector spinae plane block will be performed using an ultrasound machine with a high frequency linear probe. The patients will be in sitting position to perform the block, the skin is sterilized and the transducer will be placed across the T7 spinous process then move laterally to identify transverse process of T7. Thereafter, the probe will be moved to a parasagittal plane to visualize skin and subcutaneous tissue layers, trapezius muscle, and lastly the erector spinae muscle just superficial to the transverse processes. The in-plane technique will be used, and the tip of the needle will be inserted in the fascial plane deep to the erector spinae muscle. After 2-3 mL of normal saline injection for hydro dissection to verify the correct needle tip placement, 30 mL of 0.25% bupivacaine will be injected deep to the erector spinae muscle. The same technique will be repeated on the contralateral side.
  Other Names: ESPB
  Arms: Erector spinae plane block group (ESPB)
Procedure: Thoracic paravertebral block — Thoracic paravertebral block will be performed using an ultrasound machine with a high frequency linear probe. The patients will be in sitting position to perform the block, the skin is sterilized and the transducer will be placed across the T7 spinous process then move laterally to identify transverse process of T7. Thereafter, the probe will be moved 3-5 cm laterally to identify the paravertebral space as the target injection site. After probe being rotated into transverse orientation, the needle will be inserted using the out-plane technique. Once the needle threads the internal intercostal membrane and arrives in the paravertebral space, 3 ml of normal saline will be injected firstly. If displacement sign of the pleura occurs, 25 ml of 0.25% bupivacaine will be then injected into the confirmed paravertebral space. The same technique will be repeated on the contralateral side.
  Other Names: TPVB
  Arms: Thoracic paravertebral block group (TPVB)

SUMMARY:
The aim of this study is to compare the efficacy of ultrasound-guided bilateral erector spinae plane block and thoracic paravertebral block on perioperative analgesic control for 24 hours postoperative and fast recovery of patients undergoing laparoscopic sleeve gastrectomy using the Visual Analogue Scale.

DETAILED DESCRIPTION:
Obesity was ranked as the 5th preventable cause of death and is associated with certain diseases as non-insulin dependent diabetes mellitus, hypertension, ischemic heart disease, hyperlipidemia, and sleep apnea. Egypt has the world's 18th highest obesity prevalence, according to the World Health Organization (WHO).

Bariatric surgery has been advocated for adults with severe obesity for weight reduction purposes and lowering the health risks linked to obesity. Laparoscopic sleeve gastrectomy (LSG) is considered an efficient approach to bariatric surgery which provides an apparent weight loss and an improved weight-related quality of life with reduced postoperative morbidity but is frequently complicated by moderate to severe pain especially in the immediate postoperative period.

The Enhanced Recovery After Surgery (ERAS) recommendations for bariatric surgery currently advocate the utilization of regional anesthesia techniques, which constitute a valuable component of opioid sparing multimodal analgesia strategies to reduce intraoperative and postoperative narcotics consumption. Poorly controlled postsurgical pain is linked to decreased quality of care, surgical complications, prolonged immobility, rehabilitation and hospitalization, development of chronic pain, higher treatment costs, and a heavy burden on the healthcare system.

In 2016, the ultrasound (US)-guided erector spinae plane block (ESPB) was first described to treat thoracic neuropathic pain. The ESPB local anesthetic injectant into the fascial plane deep to the erector spinae muscle with craniocaudal distribution has an analgesic impact on somatic and visceral pain. It causes both somatic and visceral sensory blockade via acting on the ventral and dorsal rami of spinal nerves. The ESPB can provide analgesia to abdominal operations performed at a lower thoracic vertebral level (T7 or T8). However, the main concern with the ESPB is feasibility together with the potency of the block in challenging populations, such as patients suffering from obesity.

Thoracic paravertebral block (TPVB) is a classic trunk block with definite analgesic effect for both somatic and visceral pain through injecting local anaesthetic alongside the thoracic vertebrae and close to where the spinal nerves emerge from the intervertebral foramen. It produces ipsilateral, somatic and sympathetic nerve blockade in multiple contiguous thoracic dermatomes that culminate in high-quality afferent nociceptive blockade. Despite its wide use in thoracic procedures, to date, few studies have assessed the effectiveness of Thoracic paravertebral block (TPVB) in laparoscopic abdominal surgeries in an adult population.

Both blocks could be used to effectively reduce pain intensity up to 24 hours, total opioid consumption and length of hospital stay in patients undergoing laparoscopic sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 21 to 60 years.
2. Sex: males and females
3. Patients with American Society of Anesthesiologists physical status 4.classifications II-III undergoing laparoscopic sleeve gastrectomy under general anaesthesia.

Exclusion Criteria:

1. Patient refusing to participate in the study.
2. Patients with bleeding disorders.
3. A history of relevant local anaesthetic allergy.
4. Patients with muscle diseases.
5. Evidence of local infection at site of injection.
6. Pre-existing chronic pain or cognitive dysfunction (which would impede accurate engagement with postoperative quality of recovery and analgesia assessment)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Time to first Rescue Analgesia | Postoperative pain will be assessed using Visual Analogue Scale at rest (VAS-R) and with movement (VAS-M) at 30 minutes postoperative and 2, 4, 6, 8, 12, and 24 hours after surgery and Meperidine will be given accordingly.
  25 mg IV Meperidine (Pethidine) will be given as a rescue analgesia if patients complained of postoperative pain and their Visual Analogue Scale for pain ≥ 3 and to be repeated if patients continue to complain. Time to first rescue analgesia will be recorded.
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient will be asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark defines the subject's pain. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]).

SECONDARY OUTCOMES:
mean Meperidine consumption | 24 hours postoperatively
  The total requirements of rescue analgesia (Meperidine) over the first 24 hours postoperative will be recorded as mean Meperidine consumption.
Heart rate | 24 hours postoperatively
  changes in heart rate will be recorded.
Visual Analogue Scale for pain | Postoperative pain will be assessed using Visual Analogue Scale at rest (VAS-R) and with movement (VAS-M) at 30 minutes postoperative and 2, 4, 6, 8, 12, and 24 hours after surgery.
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient will be asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark defines the subject's pain. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]).
Time to perform the block | Time needed to perform the block intraoperative before induction of general anaesthesia will be recorded.
  Time taken by the investigator to perform the block.
Time to first ambulation | 24 hours postoperatively
  The time taken by the patients to start ambulation after recovery from general anaesthesia.
Systolic, Diastolic and Mean arterial blood pressures | 24 hours postoperatively
  changes in systolic, diastolic and mean arterial blood pressure will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Farouk Kamaleldin Abdelaziz, MD, Lecturer, Principal Investigator — Faculty of Medicine, Ain Shams University
Locations (1):
- Ain shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No